CLINICAL TRIAL: NCT06851052
Title: SMS - Study of Somatic Mutations Using Genome Sequencing
Acronym: SMS
Status: Enrolling by invitation | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 182435
Record Dates: First submitted 2025-02-11; First posted 2025-02-28 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-02

CONDITIONS: Somatic Mutation
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Archival tissue, such as formalin fixed paraffin embedded samples, previously collected from the donor for clinical purposes. Other materials that may be included: Extracted DNA/RNA samples, plucked hairs and DNA or cells extracted from plucked hairs, skin biopsies of up to 4mm in diameter, urine and cells obtained from urine, blood samples and cells obtained from blood samples, tissue removed at a future, clinically indicated surgical procedure surplus to diagnostic requirements and cell lines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Controls: Healthy adults with capacity to consent these may be patient's relatives either recruited by the research nurse or clinician, or recruited via posters put up around the hospital requesting volunteers.
  Interventions: Other: sample collection; Other: Seeking consent
- Patients: Adults with capacity to consent who have been highlighted by research nurse or clinician as potentially having genetic damage caused by environmental factors, such as UV light or tobacco smoke, or other factors, such as disease history or treatments, for example radiotherapy.
  Interventions: Other: sample collection; Other: Seeking consent; Other: Sample Collection: Surgical

INTERVENTIONS:
Other: sample collection — Samples could include blood, skin biopsy, urine, plucked hair.
Other: Seeking consent
Other: Sample Collection: Surgical — Excess surgical tissue (diseased tissue or tissue being removed for a clinical reason).
  Groups: Patients

SUMMARY:
Disease and tissue aging are thought to be influenced by genetic changes, or mutations, acquired throughout life. These mutations provide clues regarding the genetic damage that occurred through the lifetime of the patient, and include mutations caused by environmental factors such as ultraviolet light from sunlight or tobacco smoke affecting the skin or internal tissues, respectively. Other mutations may occur due to errors in copying the genome as cells divide. Improvements in technologies that read the genetic code have made it possible for all or selected parts of the genetic code of a human being to be "sequenced", allowing mutations (changes in the genetic code) to be detected.

DETAILED DESCRIPTION:
In this research, samples of blood, skin biopsies, plucked hairs, urine, surplus tissue removed during future planned surgery, and archived samples removed in the past will be used. The order of DNA bases in the genetic code (sequencing) in the samples will help to understand how the number and type of cells with changes in their DNA is different in tissues depending on a person's age, their exposure to environmental agents, or other factors such as disease history or treatments such as radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Controls: Healthy adults with capacity to consent
* Patients: Adults with capacity to consent who have been highlighted by research nurse or clinician as potentially having genetic damage caused by environmental factors, such as UV light or tobacco smoke, or other factors, such as disease history or treatments, for example radiotherapy.

Exclusion Criteria:

* Adults who lack capacity to consent.
* Children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who may have genetic damage caused by environmental factors, for example, a history of exposure to relevant carcinogens, such as, a high level of sunlight or tobacco. These will be identified by recruiting clinicians and research nurses in participating hospitals.
  Control participants will either be relatives of patients identified by a research nurse or clinician, or will be recruited via poster. The posters will be placed in public and staff areas in participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2028-06-14 (Estimated); Study Completion 2028-07-14 (Estimated)

PRIMARY OUTCOMES:
The study will measure the burden of somatic mutations in tissues and how this varies between controls and patients. | 10 years
  Robust statistical methods developed at the Wellcome Trust Sanger Institute will be used to analyse and interpret human genome data. This study will use bespoke computer programmes to determine the prevalence of rare mutations in normal tissue by competing the ratio of synonymous and nonsynonymous mutations for each gene analysed.
The specific mutations in genes and their prevalence will be determined. | 10 years
  Robust statistical methods developed at the Wellcome Trust Sanger Institute will be used to analyse and interpret human genome data. This study will use bespoke computer programmes to determine the prevalence of rare mutations in normal tissue by competing the ratio of synonymous and nonsynonymous mutations for each gene analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Jones, PhD, Principal Investigator — Wellcome Sanger Institute
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom